CLINICAL TRIAL: NCT07036575
Title: Integrated Program for Promoting Visual Health and Technological Applications for Individuals With Intellectual Disabilities
Brief Title: Easy-to-Read Content Effectiveness Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202504004RINA
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Health Knowledge; Intellectual Developmental Disorder; Visual Impairment
Keywords: Easy-to-Read; intellectal disability; children; special needs; visual impairment; vision health education
MeSH Terms: conditions — Intellectual Disability; Vision Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General Health Education Group (Active Comparator): Participants in this group receive standard health education using conventional visually-based educational materials (e.g., children's book) related to eye care. A trained instructor explains each image using a structured script designed for general comprehension.
  Interventions: Behavioral: Standard Visual Health Education
- Easy-to-Read Guided Teaching Group (Experimental): Participants in this group receive health education using an Easy-to-Read version of the materials, consisting of 16 simplified images with pictorial supports and plain-language text. The instruction is delivered one-on-one by a trained educator following a scripted guide optimized for individuals with intellectual or developmental disabilities.
  Interventions: Behavioral: Easy-Read Instructor-Guided Education
- Easy-to-Read Audio Self-Learning Group (Experimental): Participants in this group receive the same Easy-to-Read materials as Arm 2, but instead of guided teaching, they are instructed to operate a voice-assisted pen device to independently play back pre-recorded audio explanations linked to each image. A researcher supervises the interaction to ensure the device is used correctly, but no additional explanation is provided.
  Interventions: Behavioral: Easy-Read Audio-Based Self-Learning

INTERVENTIONS:
Behavioral: Standard Visual Health Education — Participants receive conventional eye health education using standard visual materials, explained by an instructor.
  Arms: General Health Education Group
Behavioral: Easy-Read Instructor-Guided Education — Participants receive Easy-Read health education through 16 simplified images with instructor-guided explanation using plain language and pictorial content.
  Arms: Easy-to-Read Guided Teaching Group
Behavioral: Easy-Read Audio-Based Self-Learning — Participants use a voice-assisted pen device to self-learn Easy-Read materials (16 images) with audio explanations, without additional teacher guidance.
  Arms: Easy-to-Read Audio Self-Learning Group

SUMMARY:
Individuals with intellectual disabilities face challenges in accessing medical services and health education due to communication barriers and limited support tools. Traditional information delivery methods often fail to meet their needs, leading to unequal access to preventive care and early screening.

This integrated program aims to promote visual health among individuals with intellectual disabilities through the development and implementation of inclusive technologies. The program consists of three sub-projects:

1. Visual Health Promotion and Development of an Inclusive Information Platform for Individuals with Intellectual Disabilities - developing accessible health materials for individuals with intellectual disabilities and their families.
2. Development and Promotion of a Digital Visual Health Screening System for Individuals with Intellectual Disabilities - designed to support early detection and intervention tailored to this population.
3. Development of a Healthcare Access Platform and Assistive Technologies for Individuals with Intellectual Disabilities - reducing communication barriers during medical visits through technological support.

Previously, our team developed and tested easy-to-read (ETR) materials with adults with intellectual disabilities, focusing on medical visits, eye diseases, and eye care. Once validated, these materials are planned to be adapted into digital versions and serve as the foundation for an online platform.

To evaluate the effectiveness of ETR content, we will conduct an experimental study with 250 children and adolescents with special needs from across Taipei and New Taipei City in Taiwan. Participants will receive different types of visual health education, and outcomes will be measured by improvements in their knowledge. This study aims to validate the impact of ETR resources in reducing health information inequality and improving visual health awareness in this underserved population.

DETAILED DESCRIPTION:
We will recruit 250 children and adolescents (age 3 to under 18) with intellectual disabilities or developmental delays.

1. Pre-assessment Phase:

   At the beginning of the study, background information will be collected for each participant, including date of birth, sex, current school grade, type of disability, presence of ophthalmologic conditions, whether the participant wears glasses, and past visual acuity test results.

   To assess adaptive functioning, the Vineland Adaptive Behavior Scales (VABS) will be completed by either the special education teacher or the homeroom teacher-individuals most familiar with the participant's daily behavior. The VABS is a standardized assessment tool that employs a semi-structured interview format to evaluate adaptive behaviors, including communication, daily living skills, socialization, and motor skills. It is widely used to support the diagnosis of intellectual and developmental disabilities, autism spectrum disorder, and developmental delays.

   Following the adaptive behavior assessment, participants will undergo cognitive or developmental evaluations based on age:
   * For participants aged 3 to 6, the Mullen Scales of Early Learning (MSEL) will be administered. The MSEL is a developmentally integrated assessment system that measures cognitive ability and motor development across domains such as gross and fine motor skills, visual reception, and expressive and receptive language. It provides a reliable and efficient evaluation of early learning abilities.
   * For participants aged 6 to 17, the Wechsler Intelligence Scale for Children (WISC) will be used. The WISC is a widely recognized test of intellectual functioning that assesses a child's overall intellectual ability along with five specific cognitive domains: verbal comprehension, visual spatial, fluid reasoning, working memory, and processing speed.

   In addition, participants will undergo a visual assessment, including evaluations of visual acuities, visual field, and contrast sensitivity. To ensure baseline visual recognition ability, participants will also complete a three-picture recognition test; they must correctly identify at least two out of three images to proceed in the study.

   Considering participants' physical stamina and attention span, Phase 1 will be conducted separately in advance, taking approximately 50 minutes (one class period) to complete.
2. Pre-test Phase:

   Participants will complete a brief pre-test consisting of 8 questions assessing basic eye health knowledge. Each question has two tiers: an open-ended question worth 2 points if answered correctly, followed by a yes/no question worth 1 point if the open-ended response is incorrect. This phase will take approximately 5 minutes.
3. Instructional Phase

   Participants will be randomly assigned to one of the following three instructional groups:
   * General Health Education Instruction (Control Group): Participants in this group will receive instruction using conventional materials, such as illustrated storybooks and general health education pamphlets. Instructors will guide the session by pointing to images and explaining the accompanying text.
   * Easy-to-Read Information Instruction (Experimental Group): In this group, instructors will use an easy-to-read booklet as the primary teaching material. During the session, instructors will point to the relevant images and provide explanations based on the simplified accompanying text.
   * Self-operated Easy-to-Read Audio Information (Experimental Group): Participants in this group will also use the easy-to-read booklet. However, the content will be delivered through pre-recorded audio. Using a talking pen, participants will tap on images in the booklet to trigger the corresponding narration, allowing them to learn independently through an audio-guided format.

   Following instruction, participants will be asked to confirm their understanding of the material. If full comprehension is not achieved, the instructional session will be repeated once. Regardless of comprehension level after the second attempt, the process will conclude.
4. Post-test Phase After the instructional phase, participants will complete a 5-minute distraction task involving poker games. Immediately afterward, they will retake the same eye health knowledge test used in the pre-test. The post-test phase is expected to last approximately 10 minutes.

The pre-test, instructional and post-test phase will all be conducted on the same day. The interval between these sessions and the earlier Phase 1 assessment will not exceed one month.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 3 to under 18
* Children and adolescents with intellectual disabilities and developmental delays.
* Children and adolescents who are able to correctly identify at least two out of the three images in the pre-assessment phase.

Exclusion Criteria:

* Severe cognitive impairments, hearing impairments, speech disorders, or motor disabilities that would interfere with assessment procedures or participation in the instructional activities.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Test of basic eye health knowledge Knowledge | 3 months
  This 8-question test assesses basic eye health knowledge. Each item has two stages: an open question (2 points if correct), followed by a yes/no question (1 point if correct) if the first is incorrect. It is given before and after the health education to measure learning outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ting Tsai, Study Chair — National Taiwan University
Locations (1):
- Intellectual and developmental disability centers and related institutions, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No